CLINICAL TRIAL: NCT06384365
Title: Interaktion Von Ausgewählten Inflammationsparametern, Geschmackswahrnehmung Und Geschmackspräferenzen in Abhängigkeit Von Physischer Aktivität Und Körperzusammensetzung
Brief Title: Interaction of Inflammation, Taste Perception and Preferences As a Function of Physical Activity and Body Composition
Status: Completed | Type: Observational
Sponsor: University of Vienna (Other)
Responsible Party: Principal Investigator, Barbara Lieder, Professor and Vice Chair Department of Physiological Chemistry, University of Vienna
Other Study IDs: 706014-4
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Taste, Altered
Keywords: taste; inflammation; physical activity; sweet; preference
MeSH Terms: conditions — Dysgeusia; Inflammation; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva Urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: Healthy test subjects, BMI 18.5 - 24.99 kg/m², sporting activity per week ≤ 150 minutes
- Athlectic: BMI 18.5 - 29.99 kg/m², intensive physical activity per week > 6 h (spread over min. 3 days)
  Interventions: Behavioral: Physical activity

INTERVENTIONS:
Behavioral: Physical activity — The control and the athletic group differ in the degree of physical acitvity
  Groups: Athlectic

SUMMARY:
The aim of this study is to investigate whether differences in taste perception and preference behavior can be attributed to inflammatory processes induced by physical activity. The focus will be on sweet taste and the perception of fat. A non-invasive, observational study design will be used.

DETAILED DESCRIPTION:
This study adresses the question of whether there is a connection between low-grade inflammation caused by physical activity and a change in taste perception and preference for the sweet taste. The taste perception, preference behavior and inflammation in athletic and healthy non-athletic subjects using an observational study design is investigated.

The hypothesis is that athletic test subjects, compared to healthy, physically inactive subjects, show increased inflammation values, in the range of a low-grade inflammation, and that this results in a lower sensitivity and increased preference for sweet taste.

The primary parameters to be investigated are a possible correlation between the level of physical activity physical activity or body composition and the recognition threshold for the sweet taste as well as the preference. In addition, a correlation between the concentration of TNF-α and IL-6 in saliva sweet recognition threshold and sweet preference will be investigated.

Secondary parameters to be analyzed are the preference for fatty substances, the perception threshold for the perception threshold for the fatty taste, taste receptors in saliva for the sweet and fatty taste, the concentration of 8-epi-PGF2α in the urine as a marker for oxidative stress, and the number of fungiform papillae on the tongue are determined.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* non-smoking
* normal taste and smell perception

Exclusion Criteria:

* pregnancy or breast-feeding
* regular smokers
* regular intake of medication
* metabolic diseases that require drug therapy
* ageusia or anosmia
* alcohol or drug addiction
* intake of antibiotics within the past 2 months
* vegan diet
* viral or bacterial infection wihtin the past three weeks

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 66 healthy adult participants, devided into two groups:
  Group of athletic test subjects: BMI 18.5 - 29.99 kg/m², intensive training sessions at least 3 days a week and at least 6 h per week Group of healthy, non-athletic test subjects: BMI 18.5 - 24.99 kg/m², sporting activity ≤ 150 min per week
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Taste sensitivity | day 1
  detection threshold for sweet and fatty taste analysed using a 3-AFC test
Taste preference | day 1
  preference for sweet and fatty taste analyzed by means of a Food Frequency Questionnaire and food choices from a standardized breakfast
Body composition | day 1
  body fat percentage
Low-grade inflammation | day 1
  Concentration of interleukin 6 and tumor necrosis factor alpha in unstimulated saliva

SECONDARY OUTCOMES:
Oxidative Stress | day 1
  8-epi-PGF2α analysis in urine
fungiform papillae density | day 1
  The number of fungiform papillae in a definded area of 1 cm² at the tip of the tongue is counted after staining of the tomgue with methylene blute

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lieder, PhD, Principal Investigator — University of Vienna
Locations (1):
- Christian Doppler Laboratory for Taste Research, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No